CLINICAL TRIAL: NCT04335708
Title: Effect of the Administration of the Intracellular Content Obtained From Lactobacillus Casei CRL-431 on the Antioxidant Capacity of Breast Milk
Brief Title: Effect of Intracellular Content From Lactobacillus Casei CRL-431 on Antioxidant Capacity of Breast Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Investigación en Alimentación y Desarrollo A.C. (Other)
Responsible Party: Principal Investigator, Adrian Hernandez Mendoza, Principal Investigator, Centro de Investigación en Alimentación y Desarrollo A.C.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AHM 001
Record Dates: First submitted 2020-03-17; First posted 2020-04-06 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Mothers; Lactation
Keywords: Nursing mothers; Breast milk; Lactobacillus; intracellular content; antioxidant capacity
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Daily consumption of 5 mL of edible gel with intracellular content of Lactobacillus casei CRL-431 during 30-d
  Interventions: Dietary Supplement: Postibiotic formulation
- Placebo (Placebo Comparator): Daily consumption of 5 mL of edible gel without intracellular content of Lactobacillus casei CRL-431 during 30-d
  Interventions: Dietary Supplement: Placebo formulation

INTERVENTIONS:
Dietary Supplement: Postibiotic formulation — 5 mL daily of edible gel with intracellular content of Lactobacillus casei CRL-431
  Arms: Intervention
Dietary Supplement: Placebo formulation — 5 mL daily of edible gel without intracellular content of Lactobacillus casei CRL-431
  Arms: Placebo

SUMMARY:
The objective of the present study was to evaluate the effect of the consumption of the intracellular content of Lactobacillus casei CRL-431 on the antioxidant capacity of breast milk

DETAILED DESCRIPTION:
A double blind randomized controlled clinical study of an 30-d intervention with 16 nursing mothers was carried out to evaluate the effect of the consumption of the intracellular content of Lactobacillus casei CRL-431 on the antioxidant capacity of breast milk. Once obtained the informed consent; volunteers were ramdomized into two groups (n=8) to either receive 5 mL daily: edible gel with intracellular content of Lb. casei CRL-431 (intervention group) or edible gel without intracellular content of Lb. casei CRL-431 as control (placebo). Both gels were consumed daily. Participants were asked not to change their diet or lifestyle during the intervention. We applied intention to treat for those participants who did not have good adherence and those who withdraw the study. The outcomes between groups were analyzed using a independent samples student t-test, with P value of 0.05 or less (two sided) when there was a statistical differences. Non-parametric data were analyzed with Mann-Whitney test; using statistical software.

ELIGIBILITY:
Inclusion Criteria:

* Nursing mothers between 3 and 52 weeks of lactation

Exclusion Criteria:

* Clinical evidence of chronic disease or gastrointestinal disorders
* Structural defects in the breast (breast surgery, mammary gland hypoplasia, among others)
* Mastitis
* Cancer and/or radiotherapy
* Consumption of: antioxidant supplements, probiotics, symbiotics and/or antibiotics in the month prior to recruitment.
* Alcohol or drugs consumption

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Antioxidant activity oxygen radical absorption capacity | Change from baseline antioxidant activity oxygen radical absorption capacity at day 15
  Determination of antioxidant activity by oxygen radical absorption capacity technique in breast milk
Trolox equivalent Antioxidant capacity | Change from baseline Trolox equivalent antioxidant capacity at day 15
  Determination of Trolox equivalent antioxidant capacity in breast milk
Antioxidant activity oxygen radical absorption capacity | Change from baseline antioxidant activity oxygen radical absorption capacity at day 30
  Antioxidant activity by oxygen radical absorption capacity technique in breast milk
Trolox equivalent antioxidant capacity | Change from baseline Trolox equivalent antioxidant capacity at day 30
  Determination of Trolox equivalent antioxidant capacity in breast milk

SECONDARY OUTCOMES:
Superoxide dismutase enzyme activity | Change from baseline superoxide dismutase enzyme activity at day 15
  Determination of dismutase enzyme activity in breast milk
Glutation peroxidase enzyme activity | Change from baseline glutation peroxidase enzyme activity at day 15
  Determination of glutation peroxidase enzyme activity in breast milk
Catalase enzyme activity | Change from baseline catalase enzyme activity at day 15
  Determination of catalase enzyme activity in breast milk
Glutathione activity | Change from baseline glutathione activity at day 15
  Determination of glutathione activity in breast milk
Vitamin C | Change from baseline Vitamin C at day 15
  Determination of Vitamin C in breast milk
Malondialdehyde | Change from baseline malondialdehyde at day 15
  Determination of malondialdehyde products by the thiobarbituric acid reactive substances test in breast milk
Hydrogen peroxide | Change from baseline hydrogen peroxide at day 15
  Determination of hydrogen peroxide in breast milk
Oxidative stress index | Change from baseline oxidative stress index at day 15
  Determination of oxidative stress index in breast milk

OTHER OUTCOMES:
Superoxide dismutase enzyme activity | Change from baseline superoxide dismutase enzyme activity at day 30
  Determination of dismutase enzyme activity in breast milk
Glutation peroxidase enzyme activity | Change from baseline glutton peroxidase enzyme activity at day 30
  Determination of glutation peroxidase enzyme activity in breast milk
Catalase enzyme activity | Change from baseline catalase enzyme activity at day 30
  Determination of catalase enzyme activity in breast milk
Glutathione activity | Change from baseline Glutathione activity at day 30
  Determination of glutathione activity in breast milk
Vitamin C | Change from baseline Vitamin C at day 30
  Determination of Vitamin C in breast milk
Malondialdehyde | Change from baseline malondialdehyde at day 30
  Determination of malondialdehyde in breast milk
Hydrogen peroxide | Change from baseline superoxide dismutase enzyme activity at day 30
  Determination of hydrogen peroxide in breast milk
Oxidative stress index | Change from baseline oxidative stress index at day 30
  Determination of oxidative stress index in breast milk

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hernández-Mendoza, PhD, Principal Investigator — CENTRO DE INVESTIGACION EN ALIMENTACION Y DESARROLLO, A.C.
Locations (1):
- Centro de Investigacion En Alimentacion Y Desarrollo, A.C., Hermosillo, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: No